CLINICAL TRIAL: NCT04488640
Title: Compliance of Thyroid Fine Needle Aspiration Biopsy and Trucut Biopsy Results With Thyroid Imaging Reporting and Data System Score and Surgical Pathology
Brief Title: Compliance of Thyroid Fine Needle Aspiration Biopsy and Trucut Biopsy Results With TIRADS Score and Surgical Pathology
Acronym: TIRADS
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Sabahattin Destek, Principal Investigator, Clinical associate professor, Bezmialem Vakif University
Other Study IDs: 8131643
Record Dates: First submitted 2020-07-15; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Thyroid Nodule
Keywords: TI-RADS score; Thyroid fine needle aspiration biopsy; Thyroid core needle biopsy; Surgical pathology
MeSH Terms: conditions — Thyroid Nodule | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Thyroid biopsy preparations Thyroidectomy specimen preparations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thyroid fine needle aspiration biopsy group: A group of 760 people who had a thyroid nodule and who had a thyroid fine needle aspiration biopsy for diagnosis.
  Interventions: Procedure: Thyroid biopsy with ultrasound
- Thyroid core needle aspiration biopsy group: A patient group with 760 people who had a thyroid nodule and who had a thyroid fine needle aspiration biopsy for diagnosis and who underwent a core needle biopsy again. A total thyroidectomy was performed in 88 of these patients. Surgical pathology results, core needle results and TIRADS scores were compared.
  Interventions: Procedure: Thyroid biopsy with ultrasound

INTERVENTIONS:
Procedure: Thyroid biopsy with ultrasound — Patients with thyroid nodules who underwent ultrasound-guided core needle biopsy with a 20 gauge core needle biopsy apparatus were included in the study.
  Other Names: Total thyroidectomy

SUMMARY:
The investigators retrospectively reviewed the medical records of 760 patients with thyroid nodule biopsy and 88 patients who had thyroid surgery. The investigators evaluated patients' thyroid ultrasonography reports and determined Thyroid Imaging Reporting and Data System scores (TIRADS score: 1-Benign, 2- very low malignant) risk, 3-low risk, 4-medium risk, 5 -malignant high risk). The investigators evaluated patients 'existing thyroid fine needle aspiration biopsy (FNAB) reports and recorded the patients' cytology results (benign, malignant).

Documents of 88 patients who were included in the study and who underwent thyroidectomy were reviewed.Pathology reports of these patients were evaluated and surgical pathology was determined as benign in 58 patients and malignant in 30 patients.

Then, a statistical study was performed between the cor needle biopsy (CNB) results of these participants and the surgical pathology and TI-RADS scores.

ELIGIBILITY:
Inclusion Criteria:

* Having a thyroid nodule
* Being both a thyroid needle and a core biopsy

Exclusion Criteria:

* Child patients
* Pregnant patients
* Patients without a thyroid needle biopsy

Ages: 24 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thyroid biopsy data of 691 women and 69 men aged between 24-85 years were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the distribution of patients according to thyroid biopsy results. | 4-year results were included.
  Thyroid biopsy results (benign, malignant) will be compared with % of patients with these results. It will be analyzed statistically.
Examination of TIRADS score distribution according to thyroid biopsy results. | 4-year results were included.
  Thyroid biopsy results (benign, malignant) will be compared with the percentage of patients who fit the TIRADS score distribution (1-5). It will be analyzed statistically.
Evaluation of the compliance of TI-RADS scores with surgical pathology reports. | 4-year results were included.
  Surgical pathology results (benign, malignant) and TI-RADS scores (1 to 5) will be compared with% of patients matching the distribution (1-5). It will be analyzed statistically.
Evaluation of the distribution of thyroid biopsy results and surgical pathology results. | 4-year results were included.
  The % of patients who match the distribution of thyroid biopsy results (benign, malignant) and surgical pathology results (benign, malignant) will be compared. It will be analyzed statistically.

CONTACTS AND LOCATIONS:
Overall Officials: Beyza Benturk, Dr, Study Chair — Bezmialem Vakif University

IPD SHARING:
Plan to Share IPD: Undecided
We retrospectively analyzed the medical records of 760 patients with thyroid nodule biopsy and 88 patients who had thyroid surgery. We retrospectively analyzed the medical records of 760 patients who had undergone thyroid fine needle aspiration biopsy and core needle biopsy (CNB) and 88 patients who had thyroid surgery. After the study, core needle biopsy results were statistically compatible with Thyroid Imaging Reporting and Data System (TI-RADS) scores and surgical pathology results in patients. As a result, CNB is a reliable diagnostic method.

REFERENCES:
- [Result] Singh Ospina N, Brito JP, Maraka S, Espinosa de Ycaza AE, Rodriguez-Gutierrez R, Gionfriddo MR, Castaneda-Guarderas A, Benkhadra K, Al Nofal A, Erwin P, Morris JC, Castro MR, Montori VM. Diagnostic accuracy of ultrasound-guided fine needle aspiration biopsy for thyroid malignancy: systematic review and meta-analysis. Endocrine. 2016 Sep;53(3):651-61. doi: 10.1007/s12020-016-0921-x. Epub 2016 Apr 12. PMID 27071659
- [Result] Singaporewalla RM, Hwee J, Lang TU, Desai V. Clinico-pathological Correlation of Thyroid Nodule Ultrasound and Cytology Using the TIRADS and Bethesda Classifications. World J Surg. 2017 Jul;41(7):1807-1811. doi: 10.1007/s00268-017-3919-5. PMID 28251273
- [Result] Lew JI, Snyder RA, Sanchez YM, Solorzano CC. Fine needle aspiration of the thyroid: correlation with final histopathology in a surgical series of 797 patients. J Am Coll Surg. 2011 Jul;213(1):188-94; discussion 194-5. doi: 10.1016/j.jamcollsurg.2011.04.029. Epub 2011 May 20. PMID 21601489
- [Result] Kim SY, Lee HS, Moon J, Kim EK, Moon HJ, Yoon JH, Kwak JY. Fine-needle aspiration versus core needle biopsy for diagnosis of thyroid malignancy and neoplasm: a matched cohort study. Eur Radiol. 2017 Feb;27(2):801-811. doi: 10.1007/s00330-016-4424-1. Epub 2016 Jun 3. PMID 27260342
- [Result] Hahn SY, Shin JH, Oh YL, Park KW, Lim Y. Comparison Between Fine Needle Aspiration and Core Needle Biopsy for the Diagnosis of Thyroid Nodules: Effective Indications According to US Findings. Sci Rep. 2020 Mar 18;10(1):4969. doi: 10.1038/s41598-020-60872-z. PMID 32188891